CLINICAL TRIAL: NCT03349996
Title: Belgian Physician-initiated Trial Investigating the LifeStream Peripheral Stent Graft System for the Treatment of Complex TASC C and D Iliac Lesions
Brief Title: Belgian Trial Investigating the LifeStream Stent in Complex TASC C and D Iliac Lesions
Acronym: BELSTREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID3-20170704
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LifeStream Peripheral Stent Graft System (Experimental): Patients treated with the LifeStream Peripheral Stent Graft System
  Interventions: Device: LifeStream Peripheral Stent Graft System

INTERVENTIONS:
Device: LifeStream Peripheral Stent Graft System — Patients will be treated with the LifeStream Peripheral Stent Graft System

SUMMARY:
The BELSTREAM Trial investigates the efficacy of the LifeStream Peripheral Stent Graft System in the treatment of iliac stenotic or occlusive lesions (TASC C and D). An expected total of 70 patients will be treated. The lesion is located within the native Iliac arteries. Prior to stenting with the LifeStream Peripheral Stent Graft System, pre-dilatation can be performed according to the physician's discretion. Also post-dilatation can be performed according to the physician's discretion. Patients will be invited for a follow-up visit at 1, 6, 12, 24 ,36 ,48 and 60-month post-procedure. .The primary efficacy endpoint of the study is the primary patency at 12 months. The primary safety endpoint is the freedom of periprocedural Serious Adverse Events (SAEs). Secondary endpoint include primary patency rate at 1 ,6 ,24 ,36 ,48 and 60 month, stent graft occlusion rate at pre-discharge, 1 ,6 ,12 ,24 ,36 ,48 and 60-month follow-up, anke-brachial index (ABI) at 1 ,6 ,12 ,24 ,36 ,48 and 60-month follow-up, amputation rate at 1 ,6 ,12 ,24 ,36 ,48 and 60-month follow-up, technical success and clinical success at 1 ,6 ,12 ,24 ,36 ,48 and 60-month follow-up.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to evaluate, in a controlled setting, the long-term safety and efficacy of the LifeStream Peripheral Stent Graft System in clinical settings post CE-certification when used according to the indications of the IFU with focus on the treatment of complex TASC C and D iliac lesions.

Patients will be selected based on the investigator's assessment, evaluation of the underlying disease and the eligibility criteria. The patient's medical condition should be stable, with no underlying medical condition which would prevent them from performing the required testing or from completing the study. Patients should also be geographically stable, willing and able to cooperate in this clinical study and remain available for long-term follow-up. A patient is considered enrolled in the study after obtaining the patients informed consent, if there is full compliance with the study eligibility criteria and after successful guidewire passage through the study target lesion.

Prior to the index procedure the following tests and clinical data will be collected: informed consent for data collection, demographics, medical history, medication record, physical examination, clinical category of chronic limb ischemia (Rutherford category) and resting ankle-brachial index (ABI).

During the procedure, the vascular access can be achieved to the investigator's standard clinical practice. After successful lesion passage, diagnostic angiography of the lesion area and distal run-off is performed and angiographic measurements (vessel diameter, percentage stenosis and lesion length) are collected. At the physician's discretion, the patient receives at least 1 LifeStream Peripheral Stent Graft System. Pre- and post-dilatation are according to the physician's discretion. No other adjunctive therapies (atherectomy, laser) are allowed. The complete iliac vasculature should be treated in one single session, staged interventions are not allowed. All outflow-limiting lesions must be treated according to the hospital treatment standard.

The regular follow-ups are necessary to monitor the condition of the patient and the stent/procedure. Patients will be invited for a follow-up visit at 1 ,6 ,12 ,24 ,36 ,48 and 60-months after the index procedure. The following data will be collected during these follow-up visit: medication record, physical examination, rutherford categorization, ABI and color flow doppler ultrasound.

ELIGIBILITY:
General inclusion criteria:

* Corresponding to the CE-mark indications/contra-indications and according to the current medical guidelines for minimally invasive peripheral interventions.
* Patient presenting with a stenotic or occlusive lesion at the iliac arteries suitable for stenting (on indication for primary stenting, based on the discretion of the investigator)
* Patient presenting a score from 2 to 4 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient is eligible for treatment with the Lifestream Peripheral Stent Graft System (Bard)

Angiographic inclusion criteria

* The target lesion is either a modified TASC-II class C or D lesion with one of the listed specifications:

  * Type C lesions

    * Bilateral Common Iliac Artery occlusions
    * Bilateral External Iliac Artery stenoses 3-10 cm long not extending into the Common Femoral Artery
  * Type D lesions

    * Unilateral occlusions of both Common Iliac and External Iliac Artery
    * Diffuse disease involving the aorta bifurcation
    * Bilateral occlusions of External Iliac Artery
* The target lesion has angiographic evidence of stenosis or restenosis post percutaneous transluminal angioplasty (PTA) > 50% or occlusion which can be passed with standard guidewire manipulation
* There is angiographic evidence of a patent Common and Deep Femoral Artery

Exclusion criteria:

* PTA is technically not possible (not feasible to access the lesion or a defect with the guidewire or balloon catheter)
* Presence of an aneurysm immediately adjacent to the site of stent graft implantation
* Lesions in or adjacent to essential collaterals(s)
* Lesions in locations subject to external compression
* Heavily calcified lesions resistant to PTA
* Patients with diffuse distal disease resulting in poor stent graft outflow
* Patients with a history of coagulation disorders
* Patients with aspirin allergy or bleeding complications and patients unable or unwilling to tolerate anticoagulant/antiplatelet therapy and/or non-responders to anticoagulant/antiplatelet therapy
* Fresh thrombus formation
* Patients with known hypersensitivity to the stent material (L605) and or polytetrafluroethylene (PTFE)
* The target lesion is either a modified TASC-II class C or D lesion with aortic or common femoral lesion involvement:

  * Type C lesions

    * Unilateral External Iliac Artery stenosis extending into the Common Femoral Artery
    * Unilateral External Iliac Artery occlusion that involves the origins of the Internal Iliac and/or Common Femoral Artery
    * Heavily calcified unilateral External Iliac Artery occlusion with involvement of the Common Femoral Artery
  * Type D lesions

    * Infra-renal aortoiliac occlusion
    * Iliac stenoses in patients with an Abdominal Aortic Aneurysm (AAA) requiring treatment and not amenable to endograft placement or other lesions requiring open aortic or iliac surgery
    * Diffuse multiple stenoses involving the unilateral Common Iliac, External Iliac and Common Femoral Artery
* Previously implanted stent(s) at the same lesion site
* Reference segment diameter is not suitable for the available stent graft design
* Untreatable lesion located at the distal outflow arteries
* Use of alternative therapy (e.g. atherectomy, cutting balloon, drug coated balloon (DCB), laser, radiation therapy) as part of the index procedure
* Patients refusing treatment
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with a history of prior life-threatening contrast medium reaction
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Study Director — ID3 Medical
Locations (7):
- Belgium (7):
  - O.L.V. Hospital, Aalst
  - Z.N.A., Antwerp
  - Imelda Hospital, Bonheiden
  - A.Z. Sint-Blasius, Dendermonde
  - Z.O.L., Genk
  - Az Groeninge, Kortrijk
  - R.Z. Heilig Hart, Tienen

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LifeStream Peripheral Stent Graft System
Started | 70
Completed | 43
Not Completed | 27
Not completed — Adverse Event | 5
Not completed — Death | 12
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Arm/Group | LifeStream Peripheral Stent Graft System
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 70
Nicotine abuse [Count of Participants; unit: Participants] | 65
Hypertension [Count of Participants; unit: Participants] | 52
Hypercholesterolemia [Count of Participants; unit: Participants] | 46
Previous arterial intervention [Count of Participants; unit: Participants] | 15
Previous coronary intervention [Count of Participants; unit: Participants] | 17
Obesity [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency at 12 Months
Description: Target lesion without a hemodynamically significant stenosis on duplex ultrasound (>50%, systolic velocity ratio greater than 2.5) and with freedom from Target Lesion Revascularization (TLR) within 12 months
Time Frame: 12 months
Population: Three patients experienced loss of primary patency before completion of the 12-month follow-up period.
Measure: Number; unit: participants
Arm/Group | LifeStream Peripheral Stent Graft System
Number analyzed (Participants) | 70
participants | 3

2. Primary Outcome: Freedom From Periprocedural Serious Adverse Events (SAEs)
Description: Periprocedural SAEs as defined according to the International Organization for Standardization guidelines (ISO) 14155:2011
Time Frame: During index procedure
Population: The periprocedural SAEs that were reported were; (1) occlusion of the iliac axis after stenting, (2) target lesion dissection after predilatation, (3) balloon rupture during predilatation and (4) target vessel perforation during the procedure.
Measure: Number; unit: Serious Adverse events
Arm/Group | LifeStream Peripheral Stent Graft System
Number analyzed (Participants) | 70
Serious Adverse events | 4

3. Secondary Outcome: Primary Patency at 1 ,6 ,24 ,36 ,48 and 60- Months Post Procedure
Description: Target lesion without a hemodynamically significant stenosis on duplex ultrasound (>50%, systolic velocity ratio greater than 2.5) and with freedom from Target Lesion Revascularization (TLR)
Time Frame: 1 ,6 ,24 ,36 ,48 and 60-months post-procedure
Population: Cumulative patency loss up to 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | LifeStream Peripheral Stent Graft System
Number analyzed (Participants) | 70
Participants
  Primary patency lost at 1 month | 0
  Primary patency lost at 6 month | 1
  Primary patency lost at 24 month | 4
  Primary patency lost at 36 month | 4
  Primary patency lost at 48 month | 4
  Primary patency lost at 60 month | 7

4. Secondary Outcome: Stent Graft Occlusion Rate
Description: Occlusion of the stent graft system
Time Frame: Pre-discharge,1 ,6 ,12 ,24 ,36 ,48 and 60-month follow-up
Population: Cumulative stent graft occlusions up to 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | LifeStream Peripheral Stent Graft System
Number analyzed (Participants) | 70
Participants
  Stent occlusion at 1 month | 0
  Stent occlusion at 6 month | 1
  Stent occlusion at 12 month | 2
  Stent occlusion at 24 month | 2
  Stent occlusion at 36 month | 2
  Stent occlusion at 48 month | 2
  Stent occlusion at 60 month | 5

5. Secondary Outcome: Ankle-Brachial Index (ABI)
Description: ABI at follow-up compared with the baseline ABI
Time Frame: 1 ,6 ,12 ,24 ,36 ,48 and 60-month post-procedure
Population: Evolution of ABI relative baseline ABI
Measure: Count of Participants; unit: Participants
Arm/Group | LifeStream Peripheral Stent Graft System
Number analyzed (Participants) | 70
Participants
  1 month post-procedure: number analyzed (Participants) | 62
  1 month post-procedure: Increased ABI compared to baseline | 56
  1 month post-procedure: Same ABI as baseline | 2
  1 month post-procedure: Decreased ABI compared to baseline | 4
  6 month post-procedure: number analyzed (Participants) | 51
  6 month post-procedure: Increased ABI compared to baseline | 50
  6 month post-procedure: Same ABI as baseline | 1
  6 month post-procedure: Decreased ABI compared to baseline | 0
  12 month post-procedure: number analyzed (Participants) | 46
  12 month post-procedure: Increased ABI compared to baseline | 43
  12 month post-procedure: Same ABI as baseline | 0
  12 month post-procedure: Decreased ABI compared to baseline | 3
  36 month post-procedure: number analyzed (Participants) | 21
  36 month post-procedure: Increased ABI compared to baseline | 20
  36 month post-procedure: Same ABI as baseline | 0
  36 month post-procedure: Decreased ABI compared to baseline | 1
  48 month post-procedure: number analyzed (Participants) | 36
  48 month post-procedure: Increased ABI compared to baseline | 34
  48 month post-procedure: Same ABI as baseline | 1
  48 month post-procedure: Decreased ABI compared to baseline | 1
  60 month post-procedure: number analyzed (Participants) | 34
  60 month post-procedure: Increased ABI compared to baseline | 30
  60 month post-procedure: Same ABI as baseline | 1
  60 month post-procedure: Decreased ABI compared to baseline | 3

6. Secondary Outcome: Amputation Rate
Description: Any amputation above the knee
Time Frame: 1 ,6 ,12 ,24 ,36 ,48 and 60-months post-procedure
Population: No above the knee amputation occurred throughout the entire study.
Measure: Count of Participants; unit: Participants
Arm/Group | LifeStream Peripheral Stent Graft System
Number analyzed (Participants) | 70
Participants | 0

7. Secondary Outcome: Technical Success
Description: Ability to achieve final residual angiographic stenosis no greater than 30%
Time Frame: Index procedure
Population: All patients reached technical success.
Measure: Count of Participants; unit: Participants
Arm/Group | LifeStream Peripheral Stent Graft System
Number analyzed (Participants) | 70
Participants | 70

8. Secondary Outcome: Clinical Success
Description: Improvement of Rutherford classification (RCC) compared to the pre-procedure classification.
Time Frame: 1 ,6 ,12 ,24 ,36 ,48 and 60-months post-procedure
Population: Rutherford classification compared to the baseline measurement
Measure: Count of Participants; unit: Participants
Arm/Group | LifeStream Peripheral Stent Graft System
Number analyzed (Participants) | 70
Participants
  1 month post-procedure: number analyzed (Participants) | 69
  1 month post-procedure: Decreased RCC compared to baseline | 67
  1 month post-procedure: Same RCC compared to baseline | 2
  1 month post-procedure: Increased RCC compared to baseline | 0
  6 month post-procedure: number analyzed (Participants) | 62
  6 month post-procedure: Decreased RCC compared to baseline | 62
  6 month post-procedure: Same RCC compared to baseline | 0
  6 month post-procedure: Increased RCC compared to baseline | 0
  12 month post-procedure: number analyzed (Participants) | 58
  12 month post-procedure: Decreased RCC compared to baseline | 54
  12 month post-procedure: Same RCC compared to baseline | 4
  12 month post-procedure: Increased RCC compared to baseline | 0
  36 month post-procedure: number analyzed (Participants) | 25
  36 month post-procedure: Decreased RCC compared to baseline | 25
  36 month post-procedure: Same RCC compared to baseline | 0
  36 month post-procedure: Increased RCC compared to baseline | 0
  48 month post-procedure: number analyzed (Participants) | 41
  48 month post-procedure: Decreased RCC compared to baseline | 40
  48 month post-procedure: Same RCC compared to baseline | 1
  48 month post-procedure: Increased RCC compared to baseline | 0
  60 month post-procedure: number analyzed (Participants) | 41
  60 month post-procedure: Decreased RCC compared to baseline | 38
  60 month post-procedure: Same RCC compared to baseline | 2
  60 month post-procedure: Increased RCC compared to baseline | 1

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | LifeStream Peripheral Stent Graft System
All-Cause Mortality (participants affected / at risk) | 12/70
Serious Adverse Events (participants affected / at risk) | 38/70
Other Adverse Events (participants affected / at risk) | 28/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LifeStream Peripheral Stent Graft System (N=70)
Severe anemia causing dyspnea and malaise (Blood and lymphatic system disorders) | 1 (1)
heart failure (Cardiac disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Fatal postoperative paralytic ileus with abdominal compartment syndrome (Gastrointestinal disorders) | 1 (1)
Positive immunochemical fecal occult blood test (Gastrointestinal disorders) | 1 (1)
Colonic polyps (Gastrointestinal disorders) | 1 (1)
gastroscopy and colonoscopy (Gastrointestinal disorders) | 1 (1)
Uncomplicated diverticulitis (Gastrointestinal disorders) | 1 (1)
Fatal condition aggravated (General disorders) | 1 (1)
Acute on chronic renal insufficiency (Infections and infestations) | 1 (1)
Fatal COVID-19 respiratory failure (Infections and infestations) | 1 (1)
Right hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Cutting wound right wrist (Injury, poisoning and procedural complications) | 1 (1)
Repeated falls, cognitive decline, aspiration pneumonia, DM2, hyperthyroidism, sinus bradycardia (Nervous system disorders) | 1 (1)
Chronic lower back pain with bilateral lumboischialgia and lower limb weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Torn meniscus (Musculoskeletal and connective tissue disorders) | 1 (1)
Cartilage damage left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fatal metastatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Fatal intracranial haemorrhage with cardiorespiratory arrest (Nervous system disorders) | 1 (1)
Brain metastases resulting in epileptic insult (Nervous system disorders) | 1 (1)
Ataxia arms and legs, instability, ethylabusus (Nervous system disorders) | 1 (1)
Phatic disorder on hypoglycemia (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Urinary tract infection and nephrolithiasis (Renal and urinary disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HPV-related high-grade PIN (Infections and infestations) | 1 (1)
Claudication (Vascular disorders) | 1 (2)
Fatal hypovolemic shock secondary to dehydration and renal failure (General disorders) | 1 (1)
Fatal thromboembolic event (Vascular disorders) | 1 (1)
Perforation of right iliac artery (Injury, poisoning and procedural complications) | 1 (1)
Perforation of right iliac artery (Vascular disorders) | 13 (14)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LifeStream Peripheral Stent Graft System (N=70)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Retrosternal pain (Cardiac disorders) | 1 (1)
Cataract development (Eye disorders) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 2 (2)
Bleeding wound of the lower leg (Injury, poisoning and procedural complications) | 2 (2)
Elevated PSA (asymptomatic) (Investigations) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Neurogenic tingling in ankles (Nervous system disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 2 (2)
Occipital headache (Nervous system disorders) | 1 (1)
Sudden dizziness causing fall; no acute intracranial trauma (Nervous system disorders) | 1 (1)
Small lacunar cerebral infarcts (Nervous system disorders) | 1 (1)
Acute ethanol intoxication (Psychiatric disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Bronchial irritation after accidental hydrochloric acid inhalation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Wound inflammation (Skin and subcutaneous tissue disorders) | 1 (1)
Balloon rupture during predilatation (Surgical and medical procedures) | 1 (1)
arterial dissection (Surgical and medical procedures) | 2 (2)
Peripheral arterial stenosis (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT03349996/Prot_SAP_000.pdf